CLINICAL TRIAL: NCT06864897
Title: The 10-year Follow-up of the Delta-TT Trial: Stability of the Delta-TT Cup with Polyethylene Insert Compared to the Delta-TT Cup with Ceramic Insert.
Brief Title: The 10-year Follow-up of the Delta-TT Trial.
Acronym: RSA-10
Status: Recruiting | Type: Observational
Sponsor: JointResearch (Other)
Responsible Party: Sponsor
Other Study IDs: NL86542.100.24
Record Dates: First submitted 2025-02-25; First posted 2025-03-07 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2024-12

CONDITIONS: Hip Dislocation
MeSH Terms: conditions — Hip Dislocation | interventions — Arthroplasty, Replacement, Hip

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Polyethylene liner
  Interventions: Device: Total hip prosthesis
- Ceramic liner
  Interventions: Device: Total hip prothesis

INTERVENTIONS:
Device: Total hip prothesis — Total hip prothesis with a Delta-TT cup, H MAX S Stem and a ceramic liner
  Groups: Ceramic liner
Device: Total hip prosthesis — Total hip prosthesis with a Delta TT cup, H MAX S stem and polyethylene liner
  Groups: Polyethylene liner

SUMMARY:
This 10-year follow-up study aims to further investigate long-term migration patterns of the uncemented Delta-TT cup and H-MAX S stem, comparing outcomes between ceramic and polyethylene liners. Given the predictive value of early RSA migration patterns at the 2-year mark for identifying implants at risk of aseptic loosening, we hypothesize that the Delta-TT cup will demonstrate good stability at the 10-year postoperative mark. Besides, it is hypothesized that migration of Delta TT-cups is comparable between ceramic and polyethylene liners.

The primary objective of this study is to measure the long-term stability of the Delta TT cup, combined with either a ceramic or cross-linked polyethylene liner, by means of RSA at 10-years postoperatively.

Secondary objectives are to measure long-term stability of the H-MAX S stem, by means of RSA at 10-year postoperatively. Furthermore the study aims to measure implant survival rates and patient-reported outcomes for both the Delta-TT cup and H-MAX S stem, comparing outcomes between the ceramic and polyethylene group.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled in the initial Delta-TT trial

Exclusion Criteria:

* Patient is unable or unwilling to sign the Informed Consent specific to this study.
* Patient is unsuitable for participation in the study based on the investigator's judgement.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients enrolled in the initial Delta-TT trial are eligible for inclusion. These patients recieved a hip prothesis including a Delta-TT cup, a H-MAX S Stem and either a polyethylene or a ceramic Liner.
Sampling Method: Probability Sample
Enrollment: 51 (Estimated)
Dates: Start 2024-10-10 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2029-05-01 (Estimated)

PRIMARY OUTCOMES:
Long-term (10-year) migration pattern of the Delta-TT cup compared between a ceramic and polyethylene liner. | 10 Years
  Measured in 3D translations and rotations by means of Radiostereometric X-ray images at 10-years postoperatively. Data will be summarized by treatment group. A mixed model analysis will be performed to assess cup migration, with liner type (polyethylene vs. ceramic) as the primary independent value. The primary outcome is the effect of the liner type on implant migration. Differences are considered significant for p-values below 0.05.

SECONDARY OUTCOMES:
Long-term (10-year) migration pattern of the H-MAX S Stem compared between a ceramic and polyethylene liner. | 10 years
  Measured in 3D translations and rotations by means of Radiostereometric X-ray images at 10-years postoperatively. Data will be summarized by treatment group. A mixed model analysis will be performed to assess stem migration, with liner type (polyethylene vs. ceramic) as the primary independent value. The primary outcome is the effect of the liner type on implant migration. Differences are considered significant for p-values below 0.05.
Implant survival of the Delta TT cup and H-MAX S stem. | 10 years
  Survival data will be collected from the Dutch Arthroplasty Register (LROI). The collected data includes: revision (yes/no), Reason for revision and survival in years. Differences in revision rates will be reported, but nog statistically tested since the study is not powered for survival analysis.
Radiographic signs of osteolysis around the Delta-TT cup. | 10 years
  Radiolucent lines are examined on lateral and anteroposterior X-rays. A radiolucent line is defined as such if the maximum width is equal to or greater than 1 mm. Orthopeadic surgeons will assess the radiolucent lines and will be blinded for liner type (obscured by researcher). Radiolucent lines are assessed in the three acetabular zones defined by DeLee and Charnley. A Chi-square test is used to compare the numer of cases with one or more radiolucent lines between the polyethylene liner group and the ceramix liner group. If there are fewer than 10 observed cases with one or more radiolucent lines in one of the two groups, the Fisher's exact test is used, which is valid for all sample sizes.
Radiographic signs of osteolysis around the H-Max S stem. | 10 years
  Radiolucent lines are examined on lateral and anteroposterior X-rays. A radiolucent line is defined as such if the maximum width is equal to or greater than 1 mm. Orthopeadic surgeons will assess the radiolucent lines and will be blinded for liner type (obscured by researcher). Radiolucent lines are assessed in the seven zones zones defined by Gruen. A Chi-square test is used to compare the numer of cases with one or more radiolucent lines between the polyethylene liner group and the ceramix liner group. If there are fewer than 10 observed cases with one or more radiolucent lines in one of the two groups, the Fisher's exact test is used, which is valid for all sample sizes.

CONTACTS AND LOCATIONS:
Overall Officials: Rudolf Poolman, PhD, Principal Investigator — Orthopedic Surgeon
Locations (1):
- OLVG Hospital, Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided